CLINICAL TRIAL: NCT00982462
Title: The Effects of Extended Duration of Long-Chain Polyunsaturated Fatty Acid (LCP)-Supplementation on Neurological and Immunological Development in Toddlers
Brief Title: Effect of Long-Chain Polyunsaturated Fatty Acid Supplementation on Toddler Cognition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Retina Foundation of the Southwest (Other)
Collaborators: DSM Nutritional Products, Inc. (Industry)
Responsible Party: Principal Investigator, Dennis Hoffman, Sr Research Scientist, Retina Foundation of the Southwest
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DSM #2009-1024
Record Dates: First submitted 2009-09-21; First posted 2009-09-23 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Infant Development
Keywords: cognition; vision; immunology; DHA; ARA; infant; nutrition
MeSH Terms: interventions — Docosahexaenoic Acids; Arachidonic Acid; Fatty Acids, Omega-3; Fatty Acids, Omega-6

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Corn oil placebo (Placebo Comparator): Micro-encapsulated powder containing corn oil placebo.
  Interventions: Dietary Supplement: Corn oil placebo
- Long-chain polyunsaturated fatty acids (Experimental): Micro-encapsulated powder containing 1:1 ratio of the omega-3 long-chain polyunsaturated fatty acids, docosahexaenoic acid (DHA) and the omega-6 fatty acid, arachidonic acid (ARA) from algal and fungal sources, respectively.
  Interventions: Dietary Supplement: Docosahexaenoic acid (DHA) and arachidonic acid (ARA)

INTERVENTIONS:
Dietary Supplement: Docosahexaenoic acid (DHA) and arachidonic acid (ARA) — Micro-encapsulated powder containing the long-chain polyunsaturated fatty acids, DHA to ARA in a 1:1 ratio. Two foil-packets containing active intervention (200mg DHA+200mg ARA) or placebo (400 mg corn oil) per day added to a selection of recommended foods.
  Other Names: Long-chain polyunsaturated fatty acids; omega-3 fatty acids; omega-6 fatty acids
  Arms: Long-chain polyunsaturated fatty acids
Dietary Supplement: Corn oil placebo — Micro-encapsulated powder containing corn oil as the placebo.
  Other Names: Long-chain polyunsaturated fatty acids; Omega-6 fatty acids
  Arms: Corn oil placebo

SUMMARY:
The hypothesis to be examined is that dietary LCP-supplementation in the second and third years of life will improve cognitive and visual maturation in early childhood.

DETAILED DESCRIPTION:
A total number of 114 toddlers at 12 months ± 2 weeks of age will be recruited and randomized to two groups (placebo or LCP-supplemented). Cognition, visual function, anthropometric, immunologic and biochemical status, and health will be assessed upon entry to evaluate equality between study groups.

The primary outcome measure for Part A will be maturation of cognition at 24 months ± 2 weeks of age (after 12 months of LCP dietary intervention) as assessed by the Bayley Scales of Infant Development (BSID)-version III. In Part B, maturation of cognition at 36 months of age (after 24 months of LCP dietary intervention) will be assessed using the Wechsler Preschool and Primary Scale of Intelligence (WPPSI-III).

The study supplements are (1) a micro-encapsulated powder containing a 1:1 ratio of the omega-3 fatty acid, docosahexaenoic acid (DHA) and the omega-6 fatty acid, arachidonic acid (ARA) from algal and fungal sources, respectively; and (2) a micro-encapsulated powder containing corn oil placebo. Two foil-packets containing either active intervention or placebo will provide 200mg DHA and 200mg ARA or 400 mg placebo oil per day to the toddler. Two packets of the powders will be added each day to a selection of recommended foods (e.g., yogurt). The duration of treatment will be from 12 to 24 months of age in Part A and in Part B will be from 24 to 36 months and followed to 42 months of age.

Secondary outcome measures are:

* COGNITION: Peabody Picture Vocabulary Test (PPVT-II; 42 mo) and the Bracken Basic Concept Scale (42 mo).
* VISION: Grating & stereoacuity (12, 24 & 36 mo); letter acuity at 36 mo.
* ANTHROPOMETRICS, HEALTH INDICES & DIETARY STATUS: Weight, height, head circumference, waist & hip measures, body mass index (BMI), skin fold fat deposition, heart rate (HR), blood pressure (BP), omega-3-targeted food questionnaire (at 12,18, 24, 30, 36, & 42 mo), childhood illnesses from birth to 36 months with emphasis on allergy and asthma chart review and a questionnaire to determine family history of asthma and allergy as well as the child's exposure to smoking (12, 24 & 36 mo).
* EXECUTIVE FUNCTION: Behavior Rating Inventory of Executive Function - Preschool Version (BRIEF-P questionnaire; 24 & 36 mo), Kansas Reflection-Impulsivity Scale for Preschoolers (KRISP; 42 mo), Dimensional Change Card Sort (DCCS; 42 mo), three Stroop Tasks (42 mo), the Grass/Snow task (42 months), and the Day/Night Task (42 months).
* SLEEP: Brief Infant Sleep Questionnaire (BSIQ;12 & 24 mo), Children's Sleep Habits Questionnaire (CSHQ; 36 & 42 mo).
* IMMUNE FUNCTION: plasma cytokine levels (12 & 24 mo), skin prick tests for specific IgEs (12 & 24 mo), plasma total IgE, salivary (secretory) IgA (12 & 24 mo), plasma C-reactive protein (CRP;12 & 24 mo).
* INDICES OF NEURAL TISSUE COMPOSITION AND COMPLIANCE: Total RBC fatty acid analysis (12 & 24 mo), buccal cheek cell phospholipids fatty acid analysis (12, 24, & 36 mo).

ELIGIBILITY:
Inclusion Criteria:

* Toddlers (12 months ± 2 weeks of age at randomization).
* Breast-fed or formula-fed during the first 12 months of life.
* Mother plans to discontinue breast-feeding/formula feeding by 13 months of age.
* Full-term at birth (37-42 weeks post-conception).
* English as the primary language in the home.

Exclusion Criteria:

* History of underlying disease or congenital malformation which, in the opinion of the Investigator, is likely to interfere with the normal growth and development of the participant or the evaluation of the participant.
* Toddler weighing <5% or >95% of the normative values in Centers for Disease Control and Prevention (CDC) growth charts released in 2000 (www.cdc.gov/growthcharts/).
* Evidence of poor food intake at time of randomization.
* Parent(s) currently supplement or plan to supplement child with >100 mg DHA per day (fish, fish oil, capsules or chewables).

Ages: 351 Days to 379 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 116 (Actual)
Dates: Start 2011-01-20 (Actual); Primary Completion 2016-06-29 (Actual); Study Completion 2016-06-29 (Actual)

PRIMARY OUTCOMES:
Maturation of cognition as assessed by the Bayley Scales of Infant Development at 24 months of age | 12 months intervention

SECONDARY OUTCOMES:
Maturation of cognition as assessed by the Wechsler Preschool and Primary Scale of Intelligence at 36 months of age | After 24 months of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Eileen E Birch, PhD, Principal Investigator — Retina Foundation of the Southwest; Dennis R Hoffman, PhD, Principal Investigator — Retina Foundation of the Southwest
Locations (1):
- Retina Foundation of the Southwest, Dallas, Texas, United States

REFERENCES:
- See also: webpage for Retina Foundation of the Southwest — http://www.retinafoundation.org